CLINICAL TRIAL: NCT00467727
Title: Lesion Characteristics' Visibility With Phase Contrast Mammography in Comparison to X-Ray Mammography for Women Undergoing X-Ray Diagnostic Mammography
Brief Title: Visibility of Lesion Characteristics With Phase Contrast Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC0702
Record Dates: First submitted 2007-04-29; First posted 2007-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Diagnostic Mammography; Breast Imaging; Phase Contrast Mammography; X-Ray Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Phase Contrast Mammography Exam
  Interventions: Other: Phase Contrast Mammography

INTERVENTIONS:
Other: Phase Contrast Mammography — Standard and magnification views

SUMMARY:
To determine if diagnostic phase contrast mammography (PCM) will provide improved image detail in assessing lesion characteristics when compared to diagnostic x-ray mammography (XM).

DETAILED DESCRIPTION:
The ability to detect lesions in mammography before they can be felt is the benefit of using this imaging modality for screening of breast cancer. Screening mammography has been proven to decrease mortality from breast cancer. Radiologists identify abnormal breast tissue in the form of microcalcifications, masses, architectural distortion, and asymmetric density by careful assessment of the characteristics of these types of lesions using the Breast Imaging Reporting and Diagnostic System (BIRADS). BIRADS was developed to provide standardization of reporting of mammographic exams. In screening mammography, while it is possible to detect lesions, often more detailed diagnostic imaging is necessary to improve the visibility of margins and edges of lesions through magnification and compression views of the lesion of interest due to spatial resolution limitations which causes geometric blurring of edges in x-ray mammography.

If the ability to clearly see margins and edges of lesions is possible at screening mammography, this would potentially decrease the overall radiation exposure currently needed to allow radiologists to be confident of their characterizations for the majority of patients using x-ray mammography. Digital mammography was developed to improve the visibility of lesions primarily in dense breasts. The reasoning was that the improved contrast range would allow for wider range of gray level differentiation but with digital mammography comes a spatial resolution limitation that blurred edges of lesions. Phase contrast mammography (PCM) was developed to improve digital mammography by providing improvement in sharpness of edges utilizing the x-ray properties of refraction.

Comparison: Phase Contrast Mammography to X-Ray Mammography for Lesion Visibility of Diagnostic Population

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years old
* Female
* Scheduled for diagnostic work-up including compression/magnification views of screening detected breast lesion

Exclusion Criteria:

* < age 40
* Male
* No screening detected findings
* Breast implants
* Any women who is pregnant or has reason to believe she is pregnant or lactating
* Women with breasts larger than the 24 x 30 cm receptor

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Measure: Lesion Visibility Comparison of Phase Contrast Mammography with X-Ray Mammography. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Etta D Pisano, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Clinical Trials, University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Tabar L, Yen MF, Vitak B, Chen HH, Smith RA, Duffy SW. Mammography service screening and mortality in breast cancer patients: 20-year follow-up before and after introduction of screening. Lancet. 2003 Apr 26;361(9367):1405-10. doi: 10.1016/S0140-6736(03)13143-1. PMID 12727392
- [Background] Tanaka T, Honda C, Matsuo S, Noma K, Oohara H, Nitta N, Ota S, Tsuchiya K, Sakashita Y, Yamada A, Yamasaki M, Furukawa A, Takahashi M, Murata K. The first trial of phase contrast imaging for digital full-field mammography using a practical molybdenum x-ray tube. Invest Radiol. 2005 Jul;40(7):385-96. doi: 10.1097/01.rli.0000165575.43381.48. PMID 15973129
- [Background] Pisano ED, Cole EB, Major S, Zong S, Hemminger BM, Muller KE, Johnston RE, Walsh R, Conant E, Fajardo LL, Feig SA, Nishikawa RM, Yaffe MJ, Williams MB, Aylward SR. Radiologists' preferences for digital mammographic display. The International Digital Mammography Development Group. Radiology. 2000 Sep;216(3):820-30. doi: 10.1148/radiology.216.3.r00se48820. PMID 10966717